CLINICAL TRIAL: NCT02883062
Title: Randomized Phase 2 Study of Neoadjuvant Chemotherapy, Carboplatin and Paclitaxel, With or Without Atezolizumab in Triple Negative Breast Cancer (TNBC)
Brief Title: Carboplatin and Paclitaxel With or Without Atezolizumab Before Surgery in Treating Patients With Newly Diagnosed, Stage II-III Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01301; NCI-2016-01301 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 201706104; 10013 (Other: Yale University Cancer Center LAO); 10013 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-08-30 (Estimated); Results first posted 2024-06-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Invasive Breast Carcinoma; Stage II Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — atezolizumab; Specimen Handling; Carboplatin; Mastectomy, Segmental; Mastectomy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (carboplatin, paclitaxel, mastectomy, lumpectomy) (Active Comparator): Patients receive carboplatin IV over 30 minutes Q3W and paclitaxel IV over 1 hour QW. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo the collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Lumpectomy; Procedure: Mastectomy; Drug: Paclitaxel
- Arm B (atezolizumab, carboplatin, paclitaxel, breast surgery) (Experimental): Patients receive atezolizumab IV over 30-60 minutes and carboplatin IV over 30 minutes Q3W, and paclitaxel IV over 1 hour QW. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo the collection of blood samples throughout the trial.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Procedure: Lumpectomy; Procedure: Mastectomy; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm B (atezolizumab, carboplatin, paclitaxel, breast surgery)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm A (carboplatin, paclitaxel, mastectomy, lumpectomy)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Lumpectomy — Undergo lumpectomy
  Other Names: Lumpectomy of Breast; Partial Mastectomy
Procedure: Mastectomy — Undergo mastectomy
  Other Names: Mammectomy
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial studies how well carboplatin and paclitaxel with or without atezolizumab before surgery works in treating patients with newly diagnosed, stage II-III triple negative breast cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving carboplatin and paclitaxel with or without atezolizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that the combination of chemotherapy and atezolizumab will increase tumor infiltrating lymphocyte (TIL) percentage compared to chemotherapy alone in patients with newly diagnosed triple negative breast cancer (TNBC) being treated with neoadjuvant chemotherapy.

II. To test the hypothesis that the combination of chemotherapy and atezolizumab will increase the pathologic complete response (pCR) rate compared to chemotherapy alone in patients with newly diagnosed TNBC being treated with neoadjuvant chemotherapy.

SECONDARY OBJECTIVE:

I. To evaluate the safety of the treatment combination of atezolizumab + carboplatin + paclitaxel.

EXPLORATORY OBJECTIVES:

I. To evaluate potential biomarkers of response to chemotherapy in combination with atezolizumab in patients with newly diagnosed TNBC.

II. To evaluate the impact of chemotherapy in combination with atezolizumab on the immune response in patients with newly diagnosed TNBC.

III. To evaluate the impact of chemotherapy in combination with atezolizumab on neoantigen-specific T cell responses in patients with newly diagnosed TNBC.

IV. To evaluate the impact of chemotherapy in combination with atezolizumab on long-term clinical endpoints such as overall survival (OS) and disease-free survival (DFS) in patients with newly diagnosed TNBC.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM A: Patients receive carboplatin intravenously (IV) over 30 minutes once every 3 weeks (Q3W) and paclitaxel IV over 1 hour once weekly (QW). Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive atezolizumab IV over 30-60 minutes and carboplatin IV over 30 minutes Q3W, and paclitaxel IV over 1 hour QW. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

In both arms, within 3-6 weeks, patients undergo mastectomy or lumpectomy. Patients also undergo the collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed new diagnosis of breast cancer
* Estrogen receptor (ER) and progesterone receptor (PR) < Allred score of 3 or =< 5% positive staining cells in the invasive component of the tumor (provided the patient is being treated as triple negative breast cancer)
* Human epidermal growth factor receptor 2 (HER2) negative by fluorescence in situ hybridization (FISH) or immunohistochemistry (IHC) staining 0 or 1+ according to National Comprehensive Cancer Network (NCCN) guidelines
* Clinical stage T2-T4c, any N, M0 primary tumor by American Joint Committee on Cancer (AJCC) 7th edition clinical staging
* Eligible for neoadjuvant chemotherapy
* No prior therapy for this disease
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 150,000/mcL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault
* International normalized ratio (INR) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Activated partial thromboplastin time (aPPT) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 180 days after the last dose of paclitaxel; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB) approved written informed consent document

Exclusion Criteria:

* Known metastatic disease
* Invasive cancer in the contralateral breast
* Patients with a previous history of non-breast malignancy are eligible only if they meet the following criteria for a cancer survivor: (1), and (2)

  * Has undergone potentially curative therapy for all prior malignancies
  * Has been considered disease-free for at least 1 year (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix)
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Treatment with any other investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia; use of bisphosphonate therapy for other reasons (e.g., osteoporosis) is allowed
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in study
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study with the exception of the planned breast cancer surgery that is part of the trial design
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Patients requiring treatment with a RANKL inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (including symptomatic sinus bradycardia), or psychiatric illness/social situations that would limit compliance with study requirements
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
* Pregnant women are excluded from this study because atezolizumab is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, breastfeeding should be discontinued if the mother is treated with atezolizumab; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2026-09-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William E Gillanders, Principal Investigator — Yale University Cancer Center LAO
Locations (14):
- United States (14):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery)
Started | 22 | 45
Completed | 16 | 45
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery) | Total
Number analyzed (Participants) | 22 | 45 | 67
Age, Continuous [Median (Full Range); unit: years] | 54 [25 to 78] | 49 [30 to 71] | 52 [25 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 45 | 67
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 22 | 42 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 11 | 13
  White | 16 | 27 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 45 | 67
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 5 | 20 | 25
  Postmenopausal | 14 | 24 | 38
  Unknown | 3 | 1 | 4
Eastern Cooperative Group (ECOG) Performance Status [Count of Participants; unit: Participants] — * ECOG 0: Fully active, able to carry on all pre-disease performance without restriction
  * ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  * ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  * ECOG 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  Participants
    0 | 21 | 41 | 62
    1 | 1 | 4 | 5
Clinical Stage [Count of Participants; unit: Participants] — * Clinical Stage II: The breast cancer is growing, but it is still contained in the breast or growth has only extended to the nearby lymph nodes.
  * Clinical Stage III: The tumor is large (more than 5 cm or about 2 inches across) or growing into nearby tissues (the skin over the breast or the muscle underneath), or the cancer has spread to many nearby lymph nodes.
  Participants
    Clinical Stage II | 14 | 31 | 45
    Clinical Stage III | 8 | 14 | 22
Nodal Involvement [Count of Participants; unit: Participants]
  Positive | 11 | 21 | 32
  Negative | 9 | 24 | 33
  Unknown | 2 | 0 | 2
Germline BRCA status [Count of Participants; unit: Participants]
  Wild type | 13 | 34 | 47
  Mutant | 4 | 5 | 9
  Unknown | 5 | 6 | 11
Baseline PD-L1 status [Count of Participants; unit: Participants]
  Negative | 5 | 19 | 24
  Positive | 4 | 16 | 20
  Unknown | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Infiltrating Lymphocyte (TIL) Percentage
Description: Will be measured by histopathologic assay. The TIL percentage after initiation of therapy will be compared between patients receiving neoadjuvant chemotherapy alone (Arm A), and patients receiving neoadjuvant chemotherapy in combination with atezolizumab (Arm B). The post-treatment TIL percentages between two arms will be summarized using descriptive statistics at each time point.
Time Frame: Baseline and between days 18-22 following completion of cycle 1 (each cycle is 3 weeks)
Population: 6 participants in Arm A were excluded. 4 of those participants withdrew consent and did not receive treatment. 2 patients did receive treatment but withdrew consent during treatment. This outcome measure is based on a modified intent-to-treat analysis (mITT). The remaining 3 participants in Arm A and 21 participants in Arm B were not evaluable because their tissue could not be evaluated or because they did not have paired samples.
Measure: Median (Full Range); unit: percentage of TIL
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery)
Number analyzed (Participants) | 13 | 24
percentage of TIL
  Baseline | 16.7 [2.5 to 75.0] | 17.5 [0.0 to 80.0]
  Days 18-22 following completion of cycle 1 | 18.3 [8.3 to 50.0] | 21.7 [3.3 to 50.0]
Statistical Analysis 1: Comparison: Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) vs Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery); Test type: Superiority; p = 0.36, Generalized estimating equation (GEE)

2. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: * Pathologic complete response rates will be summarized using contingency tables and compared using Fisher's exact test between patients receiving neoadjuvant chemotherapy alone (Arm A), and patients receiving neoadjuvant chemotherapy in combination with atezolizumab (Arm B).
  * A pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes.
Time Frame: At the time of surgery (3-6 weeks after last dose of neoadjuvant chemotherapy, neoadjuvant chemotherapy will be up to 12 weeks in length)
Population: 6 participants in Arm A were excluded. 4 of those participants withdrew consent and did not receive treatment. 2 patients did receive treatment but withdrew consent during treatment. This outcome measure is based on a modified intent-to-treat analysis (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery)
Number analyzed (Participants) | 16 | 45
Participants | 3 | 25
Statistical Analysis 1: Comparison: Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) vs Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery); Test type: Superiority; p = 0.018, Regression, Logistic

3. Secondary Outcome: Safety of the Treatment Regimen as Measured by the Number of Grade 3 or 4 Adverse Events Experienced by Participant
Description: Adverse events were classified and graded using CTCAE version 5.
Time Frame: From start of treatment of through completion of AE follow-up (median length of follow-up 2.98 months, full range 0.26-6.56 months)
Population: 4 participants in Arm A were excluded. 4 of those participants withdrew consent and did not receive treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery)
Number analyzed (Participants) | 18 | 45
Participants
  Adrenal insufficiency | 0 | 1
  ALT increase | 0 | 2
  Anemia | 2 | 8
  Anorectal infection | 0 | 1
  Arthralgia | 1 | 0
  AST increase | 0 | 1
  Diarrhea | 0 | 1
  Gastroesophageal reflux disease | 0 | 1
  Glucose intolerance | 0 | 1
  Eye inflammation | 1 | 0
  Hypocalcemia | 1 | 0
  Hypokalemia | 0 | 1
  Hypertension | 0 | 1
  Nausea | 0 | 1
  Neutropenia | 7 | 15
  Thrombocytopenia | 1 | 0
  Rash | 2 | 1
  Scleral disorder | 0 | 1
  Sepsis | 0 | 1
  Skin abscess | 0 | 2
  Syncope | 1 | 1
  Vomiting | 0 | 1
  Leukopenia | 0 | 1

4. Other Pre Specified Outcome: Incidence of Potential Biomarkers of Response
Description: Potential biomarkers include baseline TIL percentage, baseline PD-L1 expression in the tumor and tumor infiltrating immune cells, baseline immune signature, and baseline neoantigen load. Univariate and multivariate logistic regression models will be used to evaluate predictive ability of these baseline biomarkers on the response to carboplatin-based chemotherapy in combination with atezolizumab therapy. To take full advantage of such a randomized design, each model will also include the interaction term between treatment assignment and the baseline biomarker. This allows not only to answer the question whether the biomarker is predictive of pCR, but also whether the predictive ability is the same across two arms. The predictive ability will also be summarized using the area under receiver operating characteristic curves (AUC), and the 95% confidence intervals of AUC will be obtained using bootstrap resampling methods.
Time Frame: Up to the time of surgery
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Immune Response by Immune Signature
Description: The immune signature and PD-L1 expression in the tumor and tumor-infiltrating immune cells will be evaluated at baseline, after initiation of therapy (day 18-22), and at the time of surgery. The temporal changes of immune signature and PD-L1 expression in each arm will be summarized using contingency tables or descriptive statistics (means, standard deviations, medians, etc.) as appropriate. The differences of temporal change between treatment groups (Arm A versus [vs.] Arm B) or their association with clinical outcome (pCR vs. non-pCR) will also be assessed musing mixed model (PD-L1 expression) or generalized linear mixed model (immune signatures).
Time Frame: Up to the time of surgery
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Immune Response PD-L1 Expression
Description: The immune signature and PD-L1 expression in the tumor and tumor-infiltrating immune cells will be evaluated at baseline, after initiation of therapy (day 18-22), and at the time of surgery. The temporal changes of immune signature and PD-L1 expression in each arm will be summarized using contingency tables or descriptive statistics (means, standard deviations, medians, etc.) as appropriate. The differences of temporal change between treatment groups (Arm A vs. Arm B) or their association with clinical outcome (pCR vs. non-pCR) will also be assessed musing mixed model (PD-L1 expression) or generalized linear mixed model (immune signatures).
Time Frame: Up to the time of surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Neoantigen-specific T Cell Response
Description: The frequency and function of neoantigen-specific T cell across the two arms in the peripheral blood at each time point will be summarized using tools for high throughput analysis. The differences of temporal changes in neoantigen-specific T cell between treatment groups (Arm A versus Arm B) or their association with clinical outcome (pCR vs. non-pCR) will also be assessed using mixed models, followed by ad-hoc adjustment for multiple comparisons.
Time Frame: Up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Survival (OS)
Description: The distribution of OS in the two treatment arms will be described using Kaplan-Meier product limit methods and compared by log-rank tests.
Time Frame: Time from randomization to death due to any causes, assessed up to 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Disease Free Survival (DFS)
Description: The distribution of DFS in the two treatment arms will be described using Kaplan-Meier product limit methods and compared by log-rank tests.
Time Frame: Time from randomization to disease recurrence or death due to any causes, assessed up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: -Median length of follow-up was 2.98 months (full range 0.26-6.56 months). -Median length of follow-up for adverse events was 15.70 months (full range 0.03-19.61 months).
Description: -All-cause mortality was followed for all patients even if there were major protocol treatment deviations or if they did not start treatment.
Arm/Group | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery)
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/45
Serious Adverse Events (participants affected / at risk) | 4/18 | 10/45
Other Adverse Events (participants affected / at risk) | 18/18 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) (N=18) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery) (N=45)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Eye inflammation (Eye disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
ALT increase (Investigations) | 0 | 1
AST increase (Investigations) | 0 | 1
Neutropenia (Investigations) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Carboplatin, Paclitaxel, Mastectomy, Lumpectomy) (N=18) | Arm B (Atezolizumab, Carboplatin, Paclitaxel, Breast Surgery) (N=45)
Anemia (Blood and lymphatic system disorders) | 13 | 38
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Swollen right neck lymph node (Blood and lymphatic system disorders) | 0 | 1
Chest pain-cardiac (Cardiac disorders) | 1 | 1
Chest tightness (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 3
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 3
Ear drainage (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1
Aura (Eye disorders) | 0 | 1
Blurred vision (Eye disorders) | 2 | 5
Cataract (Eye disorders) | 0 | 1
Difficulty focusing (Eye disorders) | 0 | 1
Double vision (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eye spasms (Eye disorders) | 0 | 2
Eye twitching (Eye disorders) | 0 | 2
Eyelid function disorder (Eye disorders) | 1 | 1
Iritis (Eye disorders) | 0 | 1
Scleral disorder (Eye disorders) | 0 | 1
Stye in right eye (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 10
Bloating (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 8 | 22
Diarrhea (Gastrointestinal disorders) | 7 | 23
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 6
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 5
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 1
Intermittent loose stools (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 9 | 27
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Thrush (Gastrointestinal disorders) | 1 | 0
Tongue ulcer (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 9
Body aches (General disorders) | 1 | 0
Bump on left temple (General disorders) | 0 | 1
Chills (General disorders) | 0 | 3
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 1 | 6
Fatigue (General disorders) | 12 | 36
Fever (General disorders) | 1 | 7
Flu like symptoms (General disorders) | 0 | 2
Generalized itching on arms and hands (General disorders) | 1 | 0
Lightheadedness (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Night sweats (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Pain (General disorders) | 1 | 14
Allergic reaction (Immune system disorders) | 1 | 0
Bladder infection (Infections and infestations) | 0 | 1
Common cold (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 2
Mucosal infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin abscess (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 4
Yeast infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
ALT increased (Investigations) | 3 | 19
AST increased (Investigations) | 3 | 14
Alkaline phosphatase increased (Investigations) | 0 | 9
Blood bicarbonate decreased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 4 | 5
Lymphocyte count decreased (Investigations) | 3 | 17
Neutrophil count decreased (Investigations) | 11 | 29
Platelet count decreased (Investigations) | 7 | 23
Vitamin D deficiency (Investigations) | 1 | 0
Weight gain (Investigations) | 0 | 4
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 8 | 31
Anorexia (Metabolism and nutrition disorders) | 4 | 11
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 10
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 4
Hypochloremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle cramping (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Cyst cluster (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 10
Dysgeusia (Nervous system disorders) | 3 | 11
Headache (Nervous system disorders) | 4 | 16
Paresthesia (Nervous system disorders) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 15
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 5
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 2 | 10
Restlessness (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 2
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 5 | 5
Breast sensitivity (Reproductive system and breast disorders) | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 2
Libido decreased (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple deformity (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Dry nasal mucosa (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Upper respiratory irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 25
Dark spots on fingers (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Hidatadentitis suppurativa (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 4
Ingrown toenail (Skin and subcutaneous tissue disorders) | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 4
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1
PPE syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 2
Peeling lips (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 13
Red spots bilateral legs (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin plaques (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Thin/burning skin (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 3
Hematoma (Vascular disorders) | 0 | 2
Hot flashes (Vascular disorders) | 1 | 8
Hypertension (Vascular disorders) | 4 | 13
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT02883062/Prot_SAP_000.pdf